CLINICAL TRIAL: NCT06398704
Title: Investigation of the Effects of Sarcopenia and Dynapenia on Inspiratory Muscle Strength and Cardiorespiratory Fitness in Geriatric Individuals
Brief Title: Investigation of Inspiratory Muscle Strength and Cardiorespiratory Fitness in Sarcopenic Individuals
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: E-59394181-604.01-83836
Record Dates: First submitted 2024-04-28; First posted 2024-05-03 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Geriatric Individuals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sarcopenia Group: Individuals with sarcopenia according to the ISarcoPRM algorithm using the STAR method and Hand-grip
  Interventions: Other: Standart of care
- Dinapenia Group: Individuals with dynapenia according to the ISarcoPRM algorithm using the STAR method and Hand-grip
  Interventions: Other: Standart of care
- Non-sarcopenia Group: Individuals with non-sarcopenia according to the ISarcoPRM algorithm using the STAR method and Hand-grip
  Interventions: Other: Standart of care

INTERVENTIONS:
Other: Standart of care — No additional intervention was made. An evaluation was made.

SUMMARY:
The aim of our study is to examine the effects of sarcopenia and dynapenia on inspiratory muscle strength and cardiorespiratory fitness in geriatric individuals.

DETAILED DESCRIPTION:
Within the scope of the study, anterior thigh thicknesses of geriatric individuals will be evaluated by ultrasonography and individuals will be divided into 3 groups as dynapenic, sarcopenic and normal according to the ISarcoPRM algorithm, using the STAR method and Hand-grip. The Powerbreathe K5 device will be used to evaluate the inspiratory muscle strength of geriatric individuals in both groups, and the 2-minute step test will be used to evaluate cardiorespiratory fitness. The study will be carried out with 100 geriatric individuals. As a result of the study, first the inspiratory muscle strength and cardiorespiratory fitness of sarcopenic, dynapenic and non-sarcopenic groups will be compared. Afterwards, the relationship between anterior thigh thickness and inspiratory muscle strength of all geriatric individuals participating in the study will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Getting a score between 24 and 30 on the Mini Mental State Assessment
* Ability to stand without assistance for at least 90 seconds

Exclusion Criteria:

* Inability to communicate verbally
* Using a walking aid
* Older adults with severe visual impairment, neurological disorders, and/or congestive heart failure
* Older adults for whom exercise is not recommended

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric Individuals
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Ultrasonography Evaluation | Baseline
  Anterior thigh muscle thickness will be measured to evaluate sarcopenia. The obtained value will be divided by the Body Mass Index. This evaluation method is referred to in the literature as the Sonographic T-high Adjustment Rate (STAR) method. Ultrasonographic measurements will be made by a physician with at least 10 years of experience in this field using linear probes.
Evaluation of Inspiratory Muscle Strength | Baseline
  Powerbreathe K5 device was used to evaluate inspiratory muscle strength. This device is a portable, easy-to-use, accessible and reliable device used for both education and treatment purposes and evaluation purposes.
2 Minute Step Test: | Baseline
  The purpose of this test is to elevate the knees to the midpoint between the patella and the anterior-superior iliac crest. The 2 Minute Step Test is valid and reliable for assessing cardiorespiratory fitness in older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Principal Investigator — Atılım University; Özlem Yürük, Prof.Dr, Study Chair — Baskent University; Büşra Seçkinoğulları Korkusuz, MSc, Study Chair — Hacettepe University; Ferdi Yavuz, Assoc.Prof., Study Chair — European University of Lefke; Hülya Arıkan, Prof.Dr., Study Chair — Atılım University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohara DG, Pegorari MS, Oliveira Dos Santos NL, de Fatima Ribeiro Silva C, Monteiro RL, Matos AP, Jamami M. Respiratory Muscle Strength as a Discriminator of Sarcopenia in Community-Dwelling Elderly: A Cross-Sectional Study. J Nutr Health Aging. 2018;22(8):952-958. doi: 10.1007/s12603-018-1079-4. PMID 30272099
- [Background] Sawaya Y, Shiba T, Ishizaka M, Hirose T, Sato R, Kubo A, Urano T. Sarcopenia is not associated with inspiratory muscle strength but with expiratory muscle strength among older adults requiring long-term care/support. PeerJ. 2022 Feb 17;10:e12958. doi: 10.7717/peerj.12958. eCollection 2022. PMID 35194529
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253